CLINICAL TRIAL: NCT02196415
Title: Three-Dimensional Hindfoot Alignment Measurements Based On Biplanar Radiographs: Prospective Clinical Feasibility Study
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2013-0459
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-08

CONDITIONS: Congenital Medial Deviation
Keywords: Hindfoot Alignment; Rearfoot; Malalignment; biplanar radiography; 3D measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Biplanar Radiography — standard biplanar radiography of the foot
  Other Names: EOS low-dose biplanar radiography scanner

SUMMARY:
* The measurement of hindfoot alignment is a technical challenge.
* Today, hindfoot alignment is typically measured on hindfoot alignment view radiographs or long axial view radiographs. Measurements on both types of radiographs are hampered by technical shortcomings such as minimal rotational misplacement of the foot at the time of image acquisition. In previous publications our study groups demonstrated substantial measurement errors due to these shortcomings as well as bad interreader agreement.
* Hindfoot alignment measurement is feasible on MR images but hampered by the non-weight-bearing position of the patient and therefore not suited for pre-treatment evaluation.
* In an ex vivo study using plastic phantoms of a foot our research group could demonstrate superior interreader agreement and complete correction for foot misplacement at the time of image acquisition using a 3D secondary measurement technique based on biplanar low dose radiographs.
* Image acquisition using biplanar low dose radiographs is associated with a substantial reduction (about 1/7) of radiation dose applied to the patient compared to standard radiographs.
* Therefore the question arises if these excellent ex vivo results can be confirmed in a prospective clinical study.

Objectives:

1. Evaluation of technical feasibility of 3D hindfoot alignment measurements based on biplanar radiographs.
2. Reproduction of superior interreader agreement of measurements based on biplanar radiographs compared to measurements on conventional radiographs.

DETAILED DESCRIPTION:
Additional information to the brief summary:

Outcome(s): Hindfoot alignment measurement on standard radiographs and biplanar radiographs. The hindfoot angle is measured between the tibial axis and the calcaneal axis in degrees. Measurement results on plain films and based on 3D reconstructions will be compared.

Inclusion/Exclusion criteria:

* Inclusion: All patients referred for hindfoot alignment radiographs. These are all adults having suffered severe trauma or suffering from osteoarthrosis of the ankle joint. No inclusion of vulnerable participants.
* Exclusion criteria: Prior surgery, prior fracture, children and adolescents younger than the age of 20 years, known pregnancy.

Measurements and Procedures: Measurement of hindfoot alignment based on conventional radiographs and based on biplanar radiographs by two independent radiologists. Comparison of measurement results (paired-t-test, Wilcoxon signed-rank test) and calculation of interreader agreement (Intraclass correlation coefficient).

Study Product / Intervention: EOS low-dose biplanar x-ray scanner, EOS imaging, Paris, France One scan of the ankle joint to obtain an antero-posterior and lateral view.

Control Intervention: Conventional x-rays of the ankle joint (a.p., lateral, long axial or hindfoot alignment view) as referred from the clinician for treatment planning.

Number of Participants: 50 adults Based on a power analysis we think that this number of patients will enable reliable results. Because we do not know how big the differences between the measurements on standard radiographs and measurements on biplanar radiographs will be it is very difficult to perform a reasonable power analysis. In prior studies comparing torsion measurements on biplanar radiographs with CT measurements we were able to produce reliable results with the same number of patients.

Study Schedule:

First-Participant-In: June 2014 Last-Participant-Out: May 2015

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for hindfoot alignment radiographs. These are all adults having suffered severe trauma or suffering from osteoarthrosis of the ankle joint. No inclusion of vulnerable participants.

Exclusion Criteria:

* Prior surgery, prior fracture, children and adolescents younger than the age of 20 years, known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with clinically suspected hindfoot malalignment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Biplanar radiography and 3D reconstruction of hindfoot | The measurement is performed immediately after image acquisition.
  Hindfoot alignment is measured between the tibial axis and the calcaneal axis in degrees.
  Measurement on standard radiographs and biplanar radiographs are then compared.

CONTACTS AND LOCATIONS:
Overall Officials: Florian M Buck, MD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Radiology Department, Balgrist University Clinic, Zurich, Canton of Zurich, Switzerland